CLINICAL TRIAL: NCT00002045
Title: A Prospective Double-Blind Study of Retrovir in Early HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 014E; 15
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-12

CONDITIONS: HIV Infections
Keywords: Prospective Studies; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To evaluate the safety and tolerance of chronic administration of Retrovir (AZT) to adult patients with early manifestations of HIV disease. To assess the efficacy of AZT therapy in the treatment of HIV disease in these patients.

(12/01/89) Information supplied by drug company update. Study discontinued due to positive data from ACTG 016.

ELIGIBILITY:
Inclusion Criteria

Concurrent Treatment:

Allowed:

* Electron beam therapy to an area of less than 100 cm2.

Patient must have signs and symptoms of HIV infection confined to those of stages WRII-V or CDC groups III IV-A, IV-C-2 (except recurrent Salmonella bacteremia, nocardiosis, or disseminated/extrapulmonary Mycobacterium tuberculosis), and IV-E (except diffuse interstitial lymphoid pneumonitis).

* Patient must be able to give informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Evidence of nervous system dysfunction caused by factors other than HIV infection, including chronic alcohol or drug abuse.
* Present or prior known AIDS-defining opportunistic infections, lymphomas, or malignancies based on CDC criteria.
* Present or prior known systemic opportunistic diseases most recently included in the expanded CDC definition of AIDS:
* extrapulmonary or disseminated Mycobacterium tuberculosis infections, recurrent nontyphoidal Salmonella septicemia, coccidioidomycosis, diffuse interstitial lymphoid pneumonitis.
* Evidence of compromised bone marrow function defined by specified lab values.
* Evidence of HIV neurologic disease.
* Evidence of HIV-associated "wasting syndrome".
* Hypersensitivity to zidovudine (AZT).

Concurrent Medication:

Excluded:

* Cytotoxic chemotherapeutic agents.
* Steroids.
* Interferon or immunomodulating agents.
* Any antiretroviral drug including, but not limited to zidovudine (AZT), ribavirin, HPA23, AL 721, or phosphonoformate.

Patients with the following are excluded:

* Evidence of nervous system dysfunction caused by factors other than HIV infection, including chronic alcohol or drug abuse. Present or prior known AIDS-defining opportunistic infections, lymphomas, or malignancies based on CDC criteria. Present or prior known systemic opportunistic diseases most recently included in the expanded CDC definition of AIDS:
* extrapulmonary or disseminated Mycobacterium tuberculosis infections, recurrent nontyphoidal Salmonella septicemia, coccidioidomycosis, diffuse interstitial lymphoid pneumonitis.
* Evidence of compromised bone marrow function defined by specified lab values. Evidence of HIV neurologic disease.
* Evidence of HIV-associated wasting syndrome.
* Hypersensitivity to retrovir.

Prior Medication:

Excluded within 4 weeks of study entry:

* Interferon.
* Immunomodulating agents.
* Myelosuppressive drugs.
* Nephrotoxic agents.
* Other experimental chemotherapy.

Prior Treatment:

Excluded:

* Treatment with radiation therapy (with the exception of electron beam therapy to an area of less than 100 cm2).

Chronic alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States